CLINICAL TRIAL: NCT05557942
Title: A Long-Term Extension, Multi-Center Safety Study of AV-101 in Subjects With Pulmonary Arterial Hypertension (PAH) Who Have Completed Study AV-101-002 (IMPAHCT-FUL)
Brief Title: Inhaled Imatinib Pulmonary Arterial Hypertension Clinical Trial - Follow Up Long Term Extension (IMPAHCT-FUL)
Acronym: IMPAHCT-FUL
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Results from the parent study (IMPAHCT) demonstrated that while inhaled imatinib was well tolerated, it did not prove to be efficacious at any of the doses of AV-101 evaluated in the study.
Sponsor: Aerovate Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AV-101-003
Record Dates: First submitted 2022-09-15; First posted 2022-09-28 (Actual); Results first posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary Arterial Hypertension; Lungs; Pulmonary; PAH; AV-101; imatinib; IMPAHCT; IMPAHCT-FUL
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Placebo Crossover AV-101 10 mg (Experimental): Participants who previously received placebo in AV-101-002 received AV-101 (imatinib) 10 milligrams (mg) administered twice daily (BID) via dry powder inhalation.
  Interventions: Drug: AV-101
- Placebo Crossover AV-101 35 mg (Experimental): Participants who previously received placebo in AV-101-002 received AV-101 (imatinib) 35 mg administered BID via dry powder inhalation.
  Interventions: Drug: AV-101
- Placebo Crossover AV-101 70 mg (Experimental): Participants who previously received placebo in AV-101-002 received AV-101 (imatinib) 70 mg administered BID via dry powder inhalation.
  Interventions: Drug: AV-101
- Continuing AV-101 10 mg (Experimental): Participants who previously received AV-101 10 mg in AV-101-002 received AV-101 (imatinib) 10 mg administered BID via dry powder inhalation.
  Interventions: Drug: AV-101
- Continuing AV-101 35 mg (Experimental): Participants who previously received AV-101 35 mg in AV-101-002 received AV-101 (imatinib) 35 mg administered BID via dry powder inhalation.
  Interventions: Drug: AV-101
- Continuing AV-101 70 mg (Experimental): Participants who previously received AV-101 70 mg in AV-101-002 received AV-101 (imatinib) 70 mg administered BID via dry powder inhalation.
  Interventions: Drug: AV-101

INTERVENTIONS:
Drug: AV-101 — AV-101 (imatinib) administered via dry powder inhalation

SUMMARY:
IMPAHCT-FUL: Inhaled Imatinib Pulmonary Arterial Hypertension Clinical Trial - Follow Up Long Term Extension (LTE) Trial was a follow up study to establish the long-term safety of AV-101. Subjects who successfully completed the 24-week placebo-controlled parent trial (AV-101-002, NCT#05036135) were offered the opportunity to continue into this LTE study. Subjects who enrolled in the study were to receive one of three active AV-101 doses until such time as the optimal dose was selected in the parent study.

ELIGIBILITY:
Key Inclusion Criteria:

To be eligible, a participant is required to be or have:

* Consented to participate in the LTE and has successfully completed the placebo-controlled 24-week Study AV-101-002.

Key Exclusion Criteria:

Subjects meeting any of the following criteria:

* The Investigator believes that it would not be in the best interest of the subject to be included in the LTE e.g., for clinical or social reasons.
* Subjects who were not compliant with study medication in AV-101-002 as assessed by the Investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2022-11-02 (Actual); Primary Completion 2024-08-08 (Actual); Study Completion 2024-08-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (72):
- United States (16):
  - Arizona Pulmonary Specialist. LTD., Phoenix, Arizona
  - University of Arizona, Department of Medicine, Tucson, Arizona
  - UCLA/David Geffen School of Medicine-Pulmonary and Criticial Care, Los Angeles, California
  - Kaiser Permanente - Los Angeles Medical Center, Los Angeles, California
  - UC Davis Medical Center, Sacramento, California
  - University of California, San Francisco, California
  - GW Medical Faculty Associates, Washington D.C., District of Columbia
  - Mayo Clinic Florida, Jacksonville, Florida
  - Emory University, Atlanta, Georgia
  - Indiana University Health, Indianapolis, Indiana
  - Tufts Medical Center, Inc., Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Ohio State University, Columbus, Ohio
  - UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
- Argentina (5):
  - Cardiologia Palmero, Buenos Aires
  - Nexo Salud Investigación Clínica, Buenos Aires
  - Sanatorio de la Trinidad Mitre, Buenos Aires
  - Insituto Medico DAMIC, Córdoba
  - Hospital Dr. Jose Maria Cullen, Santa Fe
- Australia (4):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - The Prince Charles Hospital, Chermside, Queensland
  - The Alfred Hospital, Melbourne, Victoria
- Belgium (2):
  - Cliniques Universitaires de Bruxelles Hopital Erasme, Brussels
  - UZ Leuven, Leuven
- Canada (3):
  - University of Alberta Hospital, Edmonton, Alberta
  - London Health Science Centre, London, Ontario
  - Jewish General Hospital, Montreal, Quebec
- Centro de Investigaciones Clinicas de la Universidad Catolica, Santiago, Chile
- China (8):
  - Peking Union Medical College Hospital, Beijing
  - Chongqing Medical University - The First Affiliated Hospital, Chongqing
  - Guangdong Provincial People's Hospital, Guangdong
  - Central South University - The Second Xiangya Hospital, Hunan
  - Yanan Hospital of Kunming City, Kunming
  - Gansu Provincial People's Hospital, Lanzhou
  - Southeast University (SEU) - Zhongda Hospital, Nanjing
  - Tianjin Medical University General Hospital, Tianjin
- Instituto Neumológico del Oriente S.A., Floridablanca, Colombia
- France (3):
  - Groupement Hospitalier Sud - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Hopital Arnaud de Villeneuve, Montpellier
  - Les Hôpitaux Universitaires de Strasbourg, Strasbourg
- Germany (3):
  - Universitaetsklinikum Carl Gustav Carus TU Dresden, Dresden
  - Universitaetsklinikum Giessen und Marburg GmbH Standort Giessen, Giessen
  - Universitaetsklinikum Heidelberg, Heidelberg
- Hadassah University Hospital - Ein Kerem, Jerusalem, Israel
- Italy (6):
  - Azienda Ospedaliero Universitaria Ospedali Riuniti - Foggia, Foggia
  - Ospedale San Giuseppe - Fatebenefratelli, Milan
  - Fondazione IRCCS San Gerardo Dei Tintori, Monza
  - Istituto Mediterraneo per i Trapianti e Terapie ad Alta Specializzazione, Palermo
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Azienda Ospedaliera Universitaria Policlinico Umberto I, Rome
- Pauls Stradins Clinical University Hospital, Riga, Latvia
- Mexico (2):
  - CICUM San Miguel, Guadalajara, Jalisco
  - Unidad de Investigacion Clinica en Medicina S.C., Monterrey, Nuevo León
- Poland (3):
  - Krakowski Szpital Specjalistyczny im. Jana Pawla II, Krakow
  - Wojewódzki Specjalistyczny Szpital im. Dr. Wł. Biegańskiego w Łodzi, Lodz
  - Szpital Kliniczny Przemienienia Pańskiego UM im. Marcinkowskiego, Poznan
- Portugal (2):
  - Hospital Garcia de Orta, EPE, Almada
  - Hospital Pulido Valente, Lisbon
- Singapore (2):
  - National University Hospital, Singapore
  - Tan Tock Seng Hospital, Singapore
- Center of Chest Disease Johannesburg, Johannesburg, South Africa
- Spain (7):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hosp. Universitario Gran Canaria Doctor Negrin, Las Palmas de Gran Canaria
  - Hospital 12 de Octubre, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital universtario de Salamanca, Salamanca
  - Hosp. Universitario Marques de Valdecilla, Santander
  - Hospital Universitario de Toledo, Toledo
- Imperial College Healthcare NHS Trust, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo Crossover AV-101 10 mg | Placebo Crossover AV-101 35 mg | Placebo Crossover AV-101 70 mg | Continuing AV-101 10 mg | Continuing AV-101 35 mg | Continuing AV-101 70 mg
Started | 18 | 18 | 16 | 45 | 48 | 41
Received at Least 1 Dose of Study Drug | 18 | 18 | 16 | 45 | 48 | 41
Completed ("Completed" refers to participants who completed the study) | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 18 | 18 | 16 | 45 | 48 | 41
Not completed — Death | 0 | 0 | 0 | 2 | 1 | 1
Not completed — Physician Decision | 1 | 1 | 2 | 3 | 0 | 2
Not completed — Study terminated by sponsor | 17 | 17 | 14 | 40 | 45 | 37
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: The Intent-to-treat (ITT) analysis set included all randomized participants.
Groups:
- Placebo Crossover AV-101 10 mg: Participants who previously received placebo in AV-101-002 received AV-101 (imatinib) 10 mg administered BID via dry powder inhalation.
- Total: Total of all reporting groups
Arm/Group | Placebo Crossover AV-101 10 mg | Placebo Crossover AV-101 35 mg | Placebo Crossover AV-101 70 mg | Continuing AV-101 10 mg | Continuing AV-101 35 mg | Continuing AV-101 70 mg | Total
Number analyzed (Participants) | 18 | 18 | 16 | 45 | 48 | 41 | 186
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.1 (12.45) | 45.9 (13.17) | 47.9 (11.02) | 45.5 (12.70) | 47.4 (13.98) | 46.4 (12.80) | 46.8 (12.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 13 | 34 | 38 | 35 | 150
  Male | 3 | 3 | 3 | 11 | 10 | 6 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 3 | 8 | 10 | 12 | 39
  Not Hispanic or Latino | 14 | 14 | 12 | 31 | 34 | 27 | 132
  Unknown or Not Reported | 1 | 1 | 1 | 6 | 4 | 2 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 2 | 3
  Asian | 2 | 8 | 3 | 11 | 12 | 9 | 45
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 2 | 1 | 3 | 8
  White | 15 | 8 | 11 | 27 | 31 | 24 | 116
  More than one race | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 0 | 5 | 4 | 3 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events
Description: An Adverse Event (AE) was defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious Adverse Events (SAEs) were defined as death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized participant and required medical intervention to prevent 1 of the outcomes listed in this definition. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: From date of first dose to 30 days after date of last dose (up to approximately 21 months)
Population: The Safety Analysis Set included all participants that received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Crossover AV-101 10 mg | Placebo Crossover AV-101 35 mg | Placebo Crossover AV-101 70 mg | Continuing AV-101 10 mg | Continuing AV-101 35 mg | Continuing AV-101 70 mg
Number analyzed (Participants) | 18 | 18 | 16 | 45 | 48 | 41
Participants | 9 | 11 | 12 | 26 | 25 | 21

ADVERSE EVENTS:
Time Frame: From date of first dose to date of last dose plus 30 days (up to approximately 21 months)
Description: The safety analysis set included all participants who received at least one dose of study drug.
Arm/Group | Placebo Crossover AV-101 10 mg | Placebo Crossover AV-101 35 mg | Placebo Crossover AV-101 70 mg | Continuing AV-101 10 mg | Continuing AV-101 35 mg | Continuing AV-101 70 mg
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18 | 0/16 | 2/45 | 1/48 | 1/41
Serious Adverse Events (participants affected / at risk) | 3/18 | 4/18 | 6/16 | 12/45 | 9/48 | 7/41
Other Adverse Events (participants affected / at risk) | 8/18 | 11/18 | 10/16 | 17/45 | 19/48 | 15/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Crossover AV-101 10 mg (N=18) | Placebo Crossover AV-101 35 mg (N=18) | Placebo Crossover AV-101 70 mg (N=16) | Continuing AV-101 10 mg (N=45) | Continuing AV-101 35 mg (N=48) | Continuing AV-101 70 mg (N=41)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Right ventricular failure (Cardiac disorders) | 1 | 0 | 0 | 3 | 2 | 2
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Catheter site haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1 | 2 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 2 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Atypical pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Perineal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Vascular device infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Bone lesion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 1
Device breakage (Product Issues) | 0 | 0 | 0 | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Lung hernia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Crossover AV-101 10 mg (N=18) | Placebo Crossover AV-101 35 mg (N=18) | Placebo Crossover AV-101 70 mg (N=16) | Continuing AV-101 10 mg (N=45) | Continuing AV-101 35 mg (N=48) | Continuing AV-101 70 mg (N=41)
Viral upper respiratory tract infection (Infections and infestations) | 2 | 2 | 1 | 0 | 3 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 0 | 1 | 0 | 4
COVID-19 (Infections and infestations) | 0 | 1 | 0 | 0 | 2 | 3
Influenza (Infections and infestations) | 0 | 1 | 0 | 2 | 2 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 1 | 0 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 2 | 0 | 1 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0
Atypical pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Bronchitis bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Otitis media acute (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Serratia sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Transmission of an infectious agent via transplant (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 7 | 2 | 4 | 2
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 2 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 1 | 2 | 1 | 4
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 3 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gastric disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 2 | 0 | 5 | 2 | 3
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 3 | 0 | 0 | 0
Metabolic encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 1 | 1 | 2
Fatigue (General disorders) | 2 | 0 | 0 | 1 | 1 | 0
Chest discomfort (General disorders) | 2 | 0 | 0 | 0 | 0 | 0
Catheter site haemorrhage (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Infusion site reaction (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0
Brain natriuretic peptide increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0
Oxygen saturation decreased (Investigations) | 0 | 2 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0
Blood glucose decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Blood uric acid increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Forced expiratory volume decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Glomerular filtration rate decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Heart rate increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 1 | 1 | 0
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2 | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0 | 0
Blood loss anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 1 | 2 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 2 | 0 | 0 | 0 | 0
Pulmonary valve incompetence (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0
Complications of transplanted lung (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Incision site pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Transplant dysfunction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 1 | 0
Liver injury (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Bladder irritation (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-08): https://cdn.clinicaltrials.gov/large-docs/42/NCT05557942/Prot_SAP_000.pdf